CLINICAL TRIAL: NCT04074746
Title: Bispecific NK Engager AFM13 Combined With NK Cells for Patients With Recurrent of Refractory CD30 Positive Hodgkin or Non-Hodgkin Lymphomas
Brief Title: Modified Immune Cells (AFM13-NK) and A Monoclonal Antibody (AFM13) in Treating Patients With Recurrent or Refractory CD30 Positive Hodgkin or Non-Hodgkin Lymphomas
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-1092; NCI-2019-03536 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-1092 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-06-17; First posted 2019-08-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Recurrent Anaplastic Large Cell Lymphoma; Recurrent B-Cell Non-Hodgkin Lymphoma; Recurrent Classic Hodgkin Lymphoma; Recurrent Mycosis Fungoides; Recurrent Peripheral T-Cell Lymphoma, Not Otherwise Specified; Refractory Anaplastic Large Cell Lymphoma; Refractory B-Cell Non-Hodgkin Lymphoma; Refractory Classic Hodgkin Lymphoma; Refractory Mycosis Fungoides; Refractory Peripheral T-Cell Lymphoma, Not Otherwise Specified
MeSH Terms: conditions — Lymphoma, Large-Cell, Anaplastic; Lymphoma, B-Cell; Mycosis Fungoides; Lymphoma, T-Cell | interventions — AFM13; Cyclophosphamide; fludarabine; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (AFM13-NK, AFM13) (Experimental): Patients receive standard of care fludarabine IV over 1 hour and standard of care cyclophosphamide IV over 30-60 minutes on days -5 to -3, AFM13-NK IV over 4 hours on day 0, and then AFM13 IV over 4 hours on days 7, 14, and 21.
  Interventions: Biological: Anti-CD30/CD16A Monoclonal Antibody AFM13; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Fludarabine Phosphate; Biological: Genetically Engineered Lymphocyte Therapy

INTERVENTIONS:
Biological: Anti-CD30/CD16A Monoclonal Antibody AFM13 — Given IV
  Other Names: AFM13
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
Biological: Genetically Engineered Lymphocyte Therapy — Given AFM13-NK cells IV

SUMMARY:
This phase I/II trial studies the side effects and best dose of modified umbilical cord blood immune cells (natural killer [NK] cells) combined with the antibody AFM13 (AFM13-NK) and AFM13 alone in treating patients with CD30 positive Hodgkin lymphoma or non-Hodgkin lymphoma that has come back (recurrent) or does not respond to treatment (refractory). Immunotherapy with monoclonal antibodies, such as AFM13, may help the body's immune system attack the cancer, and may interfere with the ability of cancer cells to grow and spread. Giving AFM13 loaded with NK cells followed by AFM13 alone may kill more cancer cells and decrease cancer growth in patients with CD30 positive AFM13-NK Hodgkin and Non-Hodgkin lymphomas.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To establish the safety and recommended phase II dose of umbilical cord blood (CB)-derived natural killer (NK) cells preloaded with the bispecific antibody AFM13 (AFM13-NK), followed by intravenous anti-CD30/CD16A monoclonal antibody AFM13 (AFM13) in patients with refractory/relapsed CD30-positive lymphoid malignancies based on incidence of dose limiting toxicities (DLTs) per dose level. (Phase I) II. To assess the activity of umbilical cord blood (CB)-derived natural killer (NK) cells preloaded with the bispecific antibody AFM13 (AFM13- NK), followed by intravenous AFM13 in patients with refractory/relapsed CD30-positive lymphoid malignancies. based on overall response rate (ORR), complete response (CR) rate and partial response (PR) rate. (Phase II)

SECONDARY OBJECTIVES:

I. To evaluate the duration of response. II. To evaluate the event-free survival (EFS) rate. III. To evaluate the overall survival (OS) time. IV. To quantify the persistence of infused donor CB AFM13-NK cells in the recipient.

V. To conduct comprehensive immune reconstitution studies.

OUTLINE: This is a dose-escalation study of AFM13-NK.

Patients receive standard of care fludarabine intravenously (IV) over 1 hour and standard of care cyclophosphamide IV over 30-60 minutes on days -5 to -3, AFM13-NK IV over 4 hours on day 0, and then AFM13 IV over 4 hours on days 7, 14, and 21.

After completion of study treatment, patients are followed up at 28 days, 8 weeks, 100 and 180 days and then every 3-6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of relapsed or refractory classical Hodgkin lymphoma (HL), anaplastic large cell lymphoma (ALCL), peripheral T-cell lymphoma not otherwise specified (PTCL-NOS), mycosis fungoides (MF), or B-cell non-Hodgkin lymphoma with a pre-enrollment tumor biopsy positive for CD30 by immunohistochemistry at >= 1%. Patients with HL, ALCL and MF must be refractory or intolerant to brentuximab vedotin.
* Karnofsky performance status >= 60%.
* Absolute neutrophil count >= 500/mm^3
* Platelet count >= 50,000/mm^3
* Serum creatinine clearance >= 50 ml/min, estimated using the Cockcroft-Gault equation.
* Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) =< 3 x upper limit of normal (ULN).
* Bilirubin =< 2 x ULN.
* Alkaline phosphatase (ALP) =< 2 x ULN.
* Forced expiratory volume in 1 second (FEV1) >= 50%
* Forced vital capacity (FVC) >= 50%
* Carbon monoxide diffusing capability test (DLCO) (corrected for hemoglobin [Hgb]) >= 50%
* Left ventricular ejection fraction >= 40%.
* No uncontrolled arrhythmias or symptomatic cardiac disease.
* If female of child-bearing potential, must not be pregnant or be breastfeeding and required to have a negative urine or serum pregnancy test within 3 days prior to the first dose of study drug.

  * Note: Urine pregnancy tests that cannot be confirmed as negative, require a confirmatory negative serum pregnancy test. In addition, females of childbearing potential must agree use of a highly effective method of contraception for the course of the study from 14 days prior to the first dose of study drug until 60 days after the last dose of study drug. Non-childbearing potential is defined as: Postmenopausal: defined as no menses for 12 months without an alternative medical cause. A high follicle-stimulating hormone (FSH) level in the postmenopausal range may be used to confirm post-menopausal state in women not using hormonal contraception or hormonal replacement therapy. In the absence of 12 months of amenorrhea, FSH measurements indicating post-menopausal status must be documented in patient's medical history. Permanently sterile: documented permanent sterilization e.g. hysterectomy, bilateral salpingectomy and bilateral oophorectomy. If male, surgically sterile or agrees to use a highly effective method of contraception, 14 days prior to the first dose of study drug until 60 days after the last dose of study drug.

Exclusion Criteria:

* Major surgery < 4 weeks prior to first dose of study drug.
* Any other severe or uncontrolled disease or condition which might increase the risk associated with study participation.
* Any other malignancy known to be active, with the exception of treated cervical intra-epithelial neoplasia and non-melanoma skin cancer.
* Grade >= 3 non-hematologic toxicity from prior therapy that has not resolved to grade =< 2.
* Active hepatitis B, either active carrier (hepatitis B surface antigen positive [HBsAg +]) or viremic (hepatitis B virus [HBV] deoxyribonucleic acid [DNA] >= 10,000 copies/mL, or >= 2,000 IU/mL), or hepatitis C (detectable viral load by hepatitis C virus [HCV] ribonucleic acid [RNA] polymerase chain reaction [PCR]).
* Active infection requiring parenteral antibiotics.
* Human immunodeficiency virus (HIV) infection.
* Treatment within prior 2 weeks with any anti-cancer agent, investigational or approved.
* Active central nervous system (CNS) involvement (untreated parenchymal brain metastasis or positive cytology of cerebrospinal fluid).
* Life expectancy =< 6 months.
* Previous treatment with AFM13.

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-07-18 (Actual); Primary Completion 2025-09-22 (Actual); Study Completion 2025-09-22 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 2 years
  Adverse events will be summarized by dose.

SECONDARY OUTCOMES:
Overall survival | Up to 2 years
  Distribution will be estimated using Kaplan-Meier method.
Event-free survival | Up to 2 years
  Distribution will be estimated using Kaplan-Meier method.
Overall response rate (ORR) | Up to 2 years
  Will be determined by ratio of responses over number of patients with measurable lesions. Logistic regression will be used to assess the association between ORR and disease and demographic covariates of interest.
Complete response (CR) rate | Up to 2 years
  Will be determined by ratio of CRs over number of patients with measurable lesions.
Partial response (PR) rate | Up to 2 years
  Will be determined by ratio of PRs over number of patients with measurable lesions.
Duration of response | Time of initial response to disease relapse/progression, assessed up to 2 years
Persistence of infused donor AFM13-NK cells | Up to 2 years
  Will be summarized with descriptive statistics.
Immune reconstitution studies | Up to 2 years
  Will be summarized with descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Yago L Nieto, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Nieto Y, Banerjee P, Kaur I, Basar R, Li Y, Daher M, Rafei H, Kerbauy LN, Kaplan M, Marin D, Griffin L, Barnett M, Bassett R, Uprety N, Shrestha R, Silva FR, Islam S, Ganesh C, Borneo Z, Ramdial J, Ramirez A, Hosing C, Alousi A, Popat U, Qazilbash M, Ahmed S, Iyer S, Sainz TP, Vega F, Fowlkes NW, Alexis K, Emig M, Harstrick A, Overesch A, Shpall EJ, Rezvani K. Allogeneic NK cells with a bispecific innate cell engager in refractory relapsed lymphoma: a phase 1 trial. Nat Med. 2025 Jun;31(6):1987-1993. doi: 10.1038/s41591-025-03640-8. Epub 2025 Apr 4. PMID 40186077
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2022-04-14): https://cdn.clinicaltrials.gov/large-docs/46/NCT04074746/ICF_001.pdf